CLINICAL TRIAL: NCT02646163
Title: Therapeutic Safety and Efficacy of REP 9AC (REP 2055) in HBV or HCV Infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP 101
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — REP 2055

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REP 2055 (Experimental): Treatment with REP 2055
  Interventions: Drug: REP 2055

INTERVENTIONS:
Drug: REP 2055 — (First two patients) REP 2055 is administered once weekly by slow IV infusion in dose escalation from 100 to 1200mg until a grade 3 adverse event is observed not to exceed 40 weeks of dosing.
  (Subsequent patients) 400mg of REP 2055 is administered by slow IV infusion. First week of infusion to include daily dosing followed by twice weekly dosing for 40 weeks.
  Other Names: REP 9AC

SUMMARY:
REP 9AC (REP 2055) is a nucleic acid polymer (NAP) with entry activity against hepatitis C virus and entry and post-entry antiviral activity against duck hepatitis B virus (DHBV) infection. REP 2055 has been shown to have potent prophylactic effect against HCV infection in vivo and potent therapeutic effect against established DHBV infection in vivo

The REP 101 protocol is the first-in-man proof of concept study designed to investigate the safety and antiviral activity of REP 2055 administration in human patients with chronic HBV or HCV infection.

DETAILED DESCRIPTION:
Chronic hepatitis B and C are long term conditions caused by infection of the body with the hepatitis B (HBV) and C (HCV) viruses. These infections often result in inflammation or scarring of the liver and can eventually lead to liver cirrhosis and liver failure. These infections are also one of the major causes of the development of hepatocellular carcinoma (liver cancer).

Although some drugs have been approved to treat chronic hepatitis B infections, they do not provide a complete cure except in rare cases (a cure generally means that a person loses the hepatitis B virus and develops protective surface antibodies). However, these drugs significantly decrease the risk of liver damage from the infection by slowing or stopping the virus from reproducing. Amongst the problems associated with currently available drugs are the tendency to develop resistance and the lack of clearance of the virus from the hepatocytes. There is clearly a need to identify new drugs that can benefit patients with chronic hepatitis B infections. REP 9AC is a 40mer phosphorothioate oligonucleotide that has been shown to have low toxicity and to be highly effective to treat hepatitis B infection in animals. It has been shown to be effective in protecting animal from infection and to treat animals already infected.

The efficacy of REP 9AC (REP 2055) in duck hepatitis B has been tested in collaboration with Dr. Allison Jilbert (University of Adelaide, Australia), who is a recognized expert on HBV infections. These results suggest that REP 2055 can completely eliminate the disease in a large proportion (50%) of animals following only 4 weeks of treatment. In other words, following cessation of the treatment, the viral titer does not return. If these results are replicated in humans, this will result in a paradigm shift in how patients with hepatitis B are treated. Currently available drugs can only control the disease. Once they are stopped, the viral titer returns.

This proposed study is designed to demonstrate that REP9AC can be well tolerated when given to human patients chronically infected with HBV and to evaluate if a reduction of viral titers can be observed when REP 9AC is administered as a monotherapy. Current interim data analysis from the REP 101 trial indicates the following:

1. REP 9AC is generally well tolerated at doses up to 600mg / week in all patients currently enrolled and in HBV patients at 400mg / day (for seven continuous days).
2. REP 9AC has resulted in both HBV patients achieving protective seroconversion (anti-HBs) and clearance of HBV DNA and HBsAg in their blood by 23 weeks after initiation of treatment.
3. Increasing frequency and dose of REP 9AC treatment at the start of therapy may provide more rapid seroconversion of HBV patients.
4. Increasing frequency and dose of REP 9AC treatment at the start of therapy may provide better efficacy for HCV patients.

Hepatitis C. Recent advances in the treatment of hepatitis C, using interferon and ribavirin combination therapy, have brought overall response rates to about 50% but these responses are associated with significant costs and toxicities. In view of the lack of response of many patients to standard therapy and in view of its associated toxicities, the development of new therapeutic strategies is critically important. Amphipathic polymers have been shown to have broad spectrum antiviral activities and to have very favorable pharmacokinetics in the liver making them ideal candidates for the therapy of viral hepatitis B and C.

In collaboration with Dr. Jake Liang, (Head, Liver Diseases Branch, National Institute of Health, USA), REP 9AC has been shown to provide complete protection from HCV infection in naïve animals. REP 9AC is perfectly suited for the treatment of chronic HCV infection as exposure to this drug will allow the liver to naturally eliminate infected cells by halting the continual cycle of infection of healthy liver cells. REP 9AC may eventually replace pegylated interferon and ribavirin as the standard of care owing to its activity against all genotypes of HCV and its novel mechanism of action, which does not promote the generation of drug resistance.

An entry inhibitor could be useful when used in combination therapy or could be effective as a monotherapy. This proposed study is designed to demonstrate that REP 9AC can be well tolerated when given to patients chronically infected with HCV and to evaluate if a reduction of viral titers can be observed when REP 9AC is administered as a monotherapy.

REPLICor's technology utilizes the novel properties of modified oligonucleotides (phosphorothioate oligonucleotides) as amphipathic polymers to inhibit interactions critical for viral activity. This technology is active in vitro against all known families of enveloped viruses. REPLICor's proof of concept compounds, REP 9 (REP 2006) and REP 9C (REP 2031) and its lead compound, REP 9AC (REP 2055) have also demonstrated potent antiviral activity in vivo against the following viral infections: HCV, HBV (DHBV), Cytomegalovirus, Herpes simplex virus-2, Ebola, influenza and respiratory syncytial virus.

REP 9, REP 9C and REP 9AC have been administered at therapeutically active doses in acute and chronic regimens by multiple routes of administration (parenteral, oral, topical and aerosol) in mice, rats, hamsters, guinea pigs, ducks and non human primate species with no detectable side effects. Moreover, this class of chemical compounds (phosphorothioate oligonucleotides) are known to have been well tolerated in human patients in several clinical trials.

ELIGIBILITY:
Inclusion Criteria (HBV):

* HBsAg+ for at least 6 months prior to initiation of treatment.
* HBeAg+
* HBV titer > 20000 copies/ml at start of treatment
* Treatment naïve
* HIV / hepatitis delta / HCV negative
* Compensated liver disease
* Ishak score ≤ 2
* Non cirrhotic
* No known active cytomegalovirus infection
* Willingness to utilize adequate contraception while being treated with REP 9AC (REP 2055) and for 6 months following the end of treatment
* Adequate venous access allowing weekly intravenous therapies and blood tests

Inclusion Criteria (HCV):

* HCV positive for at least 6 months prior to initiation of treatment
* Genotype 3
* HCV titer >3log IU/ml at start of treatment
* Treatment naïve
* HIV / hepatitis delta / HBV negative
* Compensated liver disease
* Chronic alanine aminotransferase or aspartate aminotransferase elevation for 6 months prior to treatment
* Ishak score ≤ 2 (patients should only have mild fibrosis)
* Non cirrhotic
* No known active cytomegalovirus infection
* Willingness to utilize adequate contraception while being treated with REP 9AC (REP 2055) and for 6 months following the end of treatment
* Adequate venous access allowing weekly intravenous therapies and blood tests

Exclusion Criteria (HBV + HCV):

* Evidence of cardiovascular disease
* Autoimmune hepatitis
* Presence of Wilson's disease
* Presence of severe NAFLD
* Evidence of any other co-existent liver disease
* Anti-nuclear antibody): positive
* Anti-HIV 1: positive
* Evidence of liver cirrhosis
* A history of ascites, hepatic encephalopathy or variceal hemorrhage
* Body weight > 100 kg
* Platelet count < 75,000, polymorphonuclear cell count < 1,500 or hematocrit < 33%
* Alfa feto protein > 100 ng/ml or the presence of a hepatic mass suggestive of hepatocellular carcinoma.
* Bilirubin > 2.5 mg/dl
* Creatinine > 1.5 mg/dl
* Platelets count < 75,000 / cmm
* Serum albumin < 35 mg/ml
* Poorly controlled diabetes mellitus
* Another serious medical disorder
* A serious psychiatric disorder
* Uncontrolled hypertension
* A history of alcohol abuse within the last year
* The use of illicit drugs within the past two years
* Inability to provide informed consent
* Positive pregnancy test
* Breastfeeding
* Inability or unwillingness to undergo a liver biopsy.
* Inability or unwillingness to provide weekly blood samples
* Poor venous access making weekly IV infusion too difficult

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of REP 2055 treatment | 40 weeks (treatment)
  To record side effects, symptoms and adverse effects of REP 2055 exposure including laboratory test abnormalities.

SECONDARY OUTCOMES:
Efficacy of REP 2055 treatment | 40 weeks (treatment) + 57 weeks (follow up)
  To assess antiviral activity of REP 2055 including serum HBsAg, HBeAg, anti-HBsAg antibodies, anti-HBeAg antibodies and HBV DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Mamun Al-Mahtab, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Farabi General Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matsumura T, Hu Z, Kato T, Dreux M, Zhang YY, Imamura M, Hiraga N, Juteau JM, Cosset FL, Chayama K, Vaillant A, Liang TJ. Amphipathic DNA polymers inhibit hepatitis C virus infection by blocking viral entry. Gastroenterology. 2009 Aug;137(2):673-81. doi: 10.1053/j.gastro.2009.04.048. Epub 2009 Apr 23. PMID 19394333
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers inhibit duck hepatitis B virus infection in vitro. Antimicrob Agents Chemother. 2013 Nov;57(11):5291-8. doi: 10.1128/AAC.01003-13. Epub 2013 Aug 12. PMID 23939902
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers prevent the establishment of duck hepatitis B virus infection in vivo. Antimicrob Agents Chemother. 2013 Nov;57(11):5299-306. doi: 10.1128/AAC.01005-13. Epub 2013 Aug 12. PMID 23939904
- [Background] Noordeen F, Scougall CA, Grosse A, Qiao Q, Ajilian BB, Reaiche-Miller G, Finnie J, Werner M, Broering R, Schlaak JF, Vaillant A, Jilbert AR. Therapeutic Antiviral Effect of the Nucleic Acid Polymer REP 2055 against Persistent Duck Hepatitis B Virus Infection. PLoS One. 2015 Nov 11;10(11):e0140909. doi: 10.1371/journal.pone.0140909. eCollection 2015. PMID 26560490
- [Derived] Al-Mahtab M, Bazinet M, Vaillant A. Safety and Efficacy of Nucleic Acid Polymers in Monotherapy and Combined with Immunotherapy in Treatment-Naive Bangladeshi Patients with HBeAg+ Chronic Hepatitis B Infection. PLoS One. 2016 Jun 3;11(6):e0156667. doi: 10.1371/journal.pone.0156667. eCollection 2016. PMID 27257978